CLINICAL TRIAL: NCT00769119
Title: A Phase II, Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy of 28 Day Oral Administration of AZD9668 in Patients With Bronchiectasis
Brief Title: A Phase II , Placebo-controlled Study to Assess Efficacy of 28 Day Oral AZD9668 in Patients With Bronchiectasis
Acronym: NEPAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0520C00010
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Results first posted 2012-07-25 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; Phase II
MeSH Terms: conditions — Bronchiectasis | interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD9668 active treatment (Experimental)
  Interventions: Drug: AZD9668
- AZD9668 placebo treatment (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9668 — 2 x 30 mg, oral tablet, twice daily for 28 days
  Arms: AZD9668 active treatment
Drug: Placebo — 2 x Matched placebo, oral tablet, twice daily for 28 days
  Arms: AZD9668 placebo treatment

SUMMARY:
The purpose of this study is to investigate if treatment with AZD9668 for 28 days is effective in treating Bronchiectasis (Brx) and if so how it compares to placebo (a substance which does not have any action).

ELIGIBILITY:
Inclusion Criteria:

* Female of non child bearing potential
* Clinical diagnosis of bronchiectasis
* Be sputum producers, with history of chronic expectoration on most days

Exclusion Criteria:

* Concomitant diagnosis of pulmonary disease other than bronchiectasis or COPD
* FEV1 of <30% of predicted normal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stockley, Prof, Principal Investigator — Queen Elizabeth Hospital, Birmingham, England; Carin Jorup, Study Director — AstraZeneca R&D Lund
Locations (9):
- Canada (5):
  - Research Site, Chemin Sainte-Foy, Quebec
  - Research Site, Calgary
  - Research Site, Montreal
  - Research Site, Ontario
  - Research Site, Vancouver
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Newcastle

REFERENCES:
- [Derived] Stockley R, De Soyza A, Gunawardena K, Perrett J, Forsman-Semb K, Entwistle N, Snell N. Phase II study of a neutrophil elastase inhibitor (AZD9668) in patients with bronchiectasis. Respir Med. 2013 Apr;107(4):524-33. doi: 10.1016/j.rmed.2012.12.009. Epub 2013 Feb 20. PMID 23433769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 25 September 2008. Last patient completed 20 April 2009. Study conducted at 6 centres in Canada and 4 centres in the UK.
Groups:
- AZD9668: AZD9668, 2 x 30 mg twice daily (bid)
- Placebo: Placebo, 2 tablets twice daily (bid)
Period: Overall Study
Arm/Group | AZD9668 | Placebo
Started | 22 | 16
Completed | 20 | 13
Not Completed | 2 | 3
Not completed — Voluntary discontinuation | 0 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Disallowed medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9668 | Placebo | Total
Number analyzed (Participants) | 22 | 16 | 38
Age Continuous [Median (Full Range); unit: years] | 61 [42 to 79] | 62 [54 to 73] | 62 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 13 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Absolute Neutrophil Count at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: The efficacy analysis set for each outcome measure includes those patients who received at least one dose of investigational product and for whom a baseline and at least one post-randomisation measurement is available for that outcome measure. Patients were analysed by to randomised treatment in accordance with the intention to treat principle.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 18 | 10
ratio | 1.08 [0.60 to 1.72] | 1.01 [0.73 to 1.60]

2. Primary Outcome: Ratio of the Percentage Neutrophil Count at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 18 | 10
ratio | 1.12 [1.02 to 1.21] | 1.04 [0.92 to 1.16]

3. Primary Outcome: 24-hour Sputum Weight(g)
Description: Sputum weight (g) collected during 24 hour periods.Change from Baseline to day 28
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 13
g | -0.15 (4.376) [lower limit 4.376] | -5.37 (3.455) [lower limit 3.455]

4. Primary Outcome: Slow Vital Capacity (SVC)
Description: Slow Vital Capacity (L) as a measure of lung function.Change from baseline to day 28
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 13
L | 0.07 (0.045) [lower limit 0.045] | -0.07 (0.057) [lower limit 0.057]

5. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced Expiratory Volume in 1 Second (L) as a measure of lung function.Change from baseline to day 28
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 13
L | 0.06 (0.021) [lower limit 0.021] | -0.04 (0.026) [lower limit 0.026]

6. Primary Outcome: Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (L) as a measure of lung function.Change from baseline to day 28
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 13
L | 0.03 (0.048) [lower limit 0.048] | 0.00 (0.061) [lower limit 0.061]

7. Primary Outcome: Forced Expiratory Flow Between 25 and 75% of Forced Vital Capacity (FEF25-75%)
Description: FEF25-75% as a measure of lung function.Change from baseline to day 28
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/s
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 13
L/s | 0.08 (0.031) [lower limit 0.031] | 0.01 (0.038) [lower limit 0.038]

8. Primary Outcome: Morning Peak Expiratory Flow (PEF)
Description: Morning Peak Expiratory Flow (L/min) as a measure of lung function.Change from mean baseline value to mean of the last 7 days on treatment
Time Frame: Last 7 days on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 21 | 16
L/min | 4.06 (6.168) [lower limit 6.168] | -4.98 (7.174) [lower limit 7.174]

9. Primary Outcome: Evening Peak Expiratory Flow (PEF)
Description: Evening Peak Expiratory Flow (L/min) as a measure of lung function.Change from mean baseline value to mean of the last 7 days on treatment
Time Frame: Last 7 days on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 21 | 16
L/min | 4.56 (6.352) [lower limit 6.352] | -1.15 (7.399) [lower limit 7.399]

10. Primary Outcome: Bronkotest Diary Card Signs and Symptoms
Description: The Bronkotest diary card includes 8 questions on signs and symptoms. Symptom scores were recorded for night-time symptoms, breathing, sputum colour, sputum amount, sputum type, wellbeing, and cough, generally scored on a scale from 0 (no symptoms) to 4 (worst symptoms). ANOVA models were fitted to compare the change from baseline between AZD9668 and placebo for each question separately, with a p-value of 0.1 considered statistically significant. The number of number of these 8 measures with significant differences is reported.
Time Frame: Last 7 days on treatment
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 21 | 16
events | 0 | 0

11. Primary Outcome: St George's Respiratory Questionnaire for COPD Patients (SGRQ-C)
Description: SGRQ total score shows the impact of COPD on patient's health status, and expressed as a percentage of impairment with scale from 0 (best health status) to 100 (worst possible status). Change from baseline to day 28.
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 19 | 13
Scores on a scale | -7.39 (3.764) [lower limit 3.764] | -1.137 (4.608) [lower limit 4.608]

12. Secondary Outcome: Ratio of Tumour Necrosis Factor Alpha (TNF α) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 12
ratio | 0.93 [0.66 to 1.30] | 1.00 [0.64 to 1.55]

13. Secondary Outcome: Ratio of Interleukin 6 (IL-6) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 12
ratio | 0.70 [0.58 to 0.86] | 0.98 [0.75 to 1.28]

14. Secondary Outcome: Ratio of Interleukin 1 Beta (IL-1β) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 11
ratio | 0.74 [0.52 to 1.07] | 0.93 [0.57 to 1.53]

15. Secondary Outcome: Ratio of Regulated on Activation, Normal T Cell Expressed and Secreted (RANTES) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 12
ratio | 0.73 [0.60 to 0.88] | 1.15 [0.90 to 1.48]

16. Secondary Outcome: Ratio of Monocyte Chemoattractant Protein-1 (MCP-1) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 12
ratio | 0.79 [0.62 to 1.01] | 1.07 [0.78 to 1.47]

17. Secondary Outcome: Ratio of Interleukin 8 (IL-8) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 12
ratio | 0.91 [0.67 to 1.23] | 1.06 [0.71 to 1.58]

18. Secondary Outcome: Ratio of Leukotriene B4 (LTB4) at End of Treatment Compared to Baseline
Description: Ratio of the mean of 3 visits at the end of the treatment period to the mean of the 3 baseline visits
Time Frame: End of treatment values from 3 visits (day 21 to 28) and baseline values from 3 visits.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 12
ratio | 0.83 [0.64 to 1.09] | 0.91 [0.64 to 1.30]

19. Secondary Outcome: Ratio of Urine Desmosine (Free) (Normalised for Creatinine) at End of Treatment Compared to Baseline
Description: Ratio of day 28 to baseline
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 12
ratio | 0.98 [0.92 to 1.05] | 0.96 [0.88 to 1.05]

20. Secondary Outcome: Ratio of Urine Desmosine (Total) (Normalised for Creatinine) at End of Treatment Compared to Baseline
Description: Ratio of day 28 to baseline
Time Frame: Baseline and day 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD9668 | Placebo
Number analyzed (Participants) | 20 | 12
ratio | 0.96 [0.83 to 1.11] | 1.05 [0.87 to 1.26]

ADVERSE EVENTS:
Arm/Group | AZD9668 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/16
Other Adverse Events (participants affected / at risk) | 13/22 | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9668 (N=22) | Placebo (N=16)
Palpitations (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Oedema Peripheral (General disorders) | 1 | 2
Chest Discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Local Swelling (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 0
Influenza (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 3
Dizziness (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 1
Depressed Mood (Psychiatric disorders) | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperaemia (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No